CLINICAL TRIAL: NCT06989411
Title: The Effectiveness Of Interferential Current Therapy On Salivary Gland Function In Individuals With Primary Sjogren's Syndrome: Single-Blind Randomized, Controlled Trial
Brief Title: Current Therapy in Primary Sjogren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, principal investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Current Therapy in pSS
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Primary Sjögren's Syndrome (pSS)

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The physiotherapist performing the evaluation was blinded to the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): treatment group
  Interventions: Other: Clinical pilates exercises +Interferential current therapy (real current)
- Group II (Placebo Comparator): Control Group
  Interventions: Other: Clinical pilates exercises+ Interferential current therapy (Placebo current)

INTERVENTIONS:
Other: Clinical pilates exercises +Interferential current therapy (real current) — All treatments were given three times a week for 8 weeks. The current intensity was determined as the mA CC level that the patient felt at the maximum but did not feel any discomfort.
  Arms: Group I
Other: Clinical pilates exercises+ Interferential current therapy (Placebo current) — All treatments were given three times a week for 8 weeks. The current intensity was set to 0.1 mA CC (necessary for the machine to work)
  Arms: Group II

SUMMARY:
Purpose:The aim of the study was to investigate the effectiveness of interferential current therapy on salivary gland function in Primary Sjogren's Syndrome (pSS).

Methods:Thirty six pSS were included in the study. Patients were randomly divided into 2 groups (Group 1 (treatment group) n=18; Group II (placebo group) n=18). Salivary flow rate measurement (SFRM), Oral Health-Related Quality of Life-United Kingdom Questionnaire (OHRQOL-UK), Oral Health Impact Profile-14 (OHIP-14), Health Assessment Questionnaire (HAQ), Beck Anxiety Inventory (BAI), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI) and Short Form-36 (SF-36) were used for evaluation. All evaluations were done pre-, posttreatment, at 3. month, at 6. month and at 9. month. Clinical pilates exercises and interferential current therapy were applied to Group I while clinical pilates exercises and interferential current therapy as placebo was applied to Group II. All treatments were given three times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with pSS according to the 2016 European League Against Rheumatism American / College of Rheumatology Classification Criteria,
* To be in the 3rd and 4th grade according to the Chisholm-Mason Grading System,
* be in the age range of 25-65 years,
* To be stable on drug use for at least 3 months or longer, (f) To have agreed to participate in the study.

Exclusion Criteria:

* To use antipsychotic, antidepressant, antihypertensive, medical agent for Parkinson's,
* Presence of viral infection,
* Presence of Diabetes Mellitus,
* Receiving head and neck radiotherapy/chemotherapy,
* Having a head and neck malignancy,
* Having undergone head and neck surgery,
* Presence of dehydration,
* Pregnancy,
* Using cigarettes and alcohol,
* Cognitive problems that affect cooperation,
* having any other disease that may affect their functions.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Salivary Flow Rate Measurement | 15 minutes
Oral Health Impact Profile-14 | 5 minutes
  Total score is between 0 and 56. A high score indicates that the quality of life related to oral and dental health decreases.
Oral Health-Related Quality of Life-United Kingdom Questionnaire | 5 minutes
  Total scores range from 16 to 80. A high score indicates that the quality of life related to oral and dental health is high.

SECONDARY OUTCOMES:
Health Assessment Questionnaire | 5 minutes
  The total score is between 0 and 3. A higher score indicates greater disability.
Beck Depression Inventory | 7 minutes
  Total summed score range of 0-63. High score means high depression
Beck Anxiety Inventory | 7 minutes
  The score range is 0-63. A high score indicates a high level of anxiety.
Short Form-36 | 10 minutes
  Each subscale has a score between 0 and 100, and a high score means the good quality of life
Pittsburgh Sleep Quality Index | 7 minutes
  Total score ranges from 0 to 21. High scores indicate poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University, Uşak, None Selected, Turkey (Türkiye)